CLINICAL TRIAL: NCT07369869
Title: Evaluating the Effects of Prebiotic and Fiber Interventions on Sleep, the Gut Microbiome, Cognition, and Stress Following 28 Days Consumption in Adults Reporting Sub-clinical Sleep Deficits: A Randomised, Double-blind, Placebo-controlled, Three-arm Parallel Groups Trial.
Brief Title: Evaluating the Effects of Prebiotic and Fiber Interventions on Sleep, the Gut Microbiome, Cognition, and Stress.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: The Coca-Cola Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 000000
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Stress; Sleep; Cognition; Nutrition; Microbiome
Keywords: sleep; gut health; cognition; stress
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Participants will be randomly allocated to consume investigational supplement (1 of 2 prebiotic/fiber 'active' compositions) for 28 days.
  Interventions: Dietary Supplement: prebiotic/fiber 'active' composition 1
- Arm 2 (Experimental): Participants will be randomly allocated to consume investigational supplement (1 of 2 prebiotic/fiber 'active' compositions) for 28 days.
  Interventions: Dietary Supplement: prebiotic/fiber 'active' composition 2
- Control (Placebo Comparator): Participants will be randomly allocated to consume control supplement for 28 days.
  Interventions: Dietary Supplement: Inactive control supplement

INTERVENTIONS:
Dietary Supplement: prebiotic/fiber 'active' composition 1 — Fiber plus micronutrients
  Arms: Arm 1
Dietary Supplement: prebiotic/fiber 'active' composition 2 — Fiber plus botanical extract
  Arms: Arm 2
Dietary Supplement: Inactive control supplement — Flavored vehicle
  Arms: Control

SUMMARY:
This will be a double-blind, placebo-controlled, parallel-group trial. Participants who are poor sleepers will be randomised to receive one of two investigational supplements, or a placebo control supplement, over a 28-day period. At baseline and following 28 days of consumption, sleep quality, gut microbiome profiles, cognitive performance, and mood will be assessed. Sleep outcome measures will also be assessed throughout the supplementation period to monitor the time course of any observed changes. A final data set of at least 66 participants is expected.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled, parallel-group trial. Participants who are poor sleepers will be randomised to receive one of two investigational supplements, or a placebo control supplement, over a 28-day period. At baseline and following 28 days of consumption, sleep quality, gut microbiome profiles, cognitive performance, and mood will be assessed. Sleep outcome measures will also be assessed throughout the supplementation period to monitor the time course of any observed changes. A final data set of at least 66 participants is expected.

Interested participants will initially be scheduled to complete a screening telephone call with the researcher. Here, electronic informed consent will first be provided by the participant, by accessing a pre-emailed link to the Qualtrics survey platform, to an account which is hosted by Northumbria University. Once consent is obtained, the participant will confirm that they do not meet any of the study exclusion criteria, and will complete the SDS-CL checklist with the researcher, over the phone. If any clinical thresholds are met, participants will be invited to a separate clinical interview (again via phonecall) with Professor Jason Ellis, employing the International Classification of Sleep Disorders (ICSD-3) criteria, to determine elligibility.

If participants progress to enrolment, they will be invited to attend a lab-based training/screening session (protocol day -7) at Northumbria University. Here, hard and wet-signed (by both the participant and the researcher) consent forms will be completed and stored on site. Participants will then be familiarised with the study protocol and procedures, including instructions on how to utilize the SleepScore and Actigraphy equipment, and how to complete the daily Sleep Diary. Participants will also be trained on the cognitive tasks. During the following 7 nights (Protocol days -7 to -1), participants will monitor their sleep via SleepScore, Actigraphy watch, and complete the daily Sleep Diary each morning. During this week, they will also drop off their pre-dose baseline stool sample at a remote drop-off location at Northumbria University.

Seven days following the lab-based screening visit (Supplement day 1, Protocol day 0), participants will attend the laboratory for their acute visit. Here, a pre-dose baseline sample of saliva and a single blood sample will be taken (for Alpha Amylase, Cortisol, Serotonin and Melatonin), and Blood Pressure, Heart Rate, Body Mass Index, and Waist-to-Hip Ratio will be measured. Participants will complete the Intake24 dietary assessment, and gastrointestinal symptoms questionnaires, as well as the Pittsburgh Sleep Quality Index (PSQI), State-Trait Anxiety Inventory (STAI), and Depression, Anxiety and Stress Scale - 21 Items (DASS-21). The cognitive task battery will additionally be completed.

After completing these measures, participants will receive instructions on the next phase of the trial. From that night, participants will consume their first dose of the investigational supplement (noting the time in their treatyment diary) 4 hours before their normal bed-time. They will monitor their sleep overnight via SleepScore, and Actigraphy watch. The following morning (supplementation day 2, protocol day 1), participants will complete their Sleep Diary. Participants will follow this procedure for the following 27 days. At some point during Protocol (Days 12-18), participants will return to Northumbria University to drop-off their interim stool sample.

On Protocol day 28, participants will return to the lab for the chronic testing visit. All of the outcome measures assessed during the acute lab visit (Protocol day 0) will be repeated here. At the end of the session, participants will be debriefed, and their participation payment arranged. At some point during Protocol (Days 27-33) participants will return to Northumbria University to drop-off their chronic stool sample.

ELIGIBILITY:
INCLUSION CRITERIA

* Participants must self-assess themselves as being in good health.
* Aged 25 to 60 years at the time of randomisation
* Fluent in English
* Identify as a 'poor sleeper' as defined subjectively (i.e. poor sleep quality, unrefreshing sleep) and a total score of >5 on the Pittsburgh Sleep Quality Index (PSQI).

EXCLUSION CRITERIA

* Member of own household currently participating in this trial
* Evidence of current or recent sleep disorders (e.g. sleep apnoea, insomnia, circadian rhythm disorders), taking any medication which exerts sedative effects, affects the CNS and/or sleep, or be currently unwell with any illness that affects sleep (i.e. disorders of the CNS). An initial screening for sleep disorders will be conducted using the Sleep Disorders Symptom Checklist-25 (SDS-CL; Klingman et al., 2017). If a participant reports positively to any of the 25 questions in terms of being affected for three nights per week, or more, this will be followed up using a clinical interview according to the International Classification of Sleep Disorders (ICSD-3) to exclude on the basis of a sleep disorder
* History of seizures or epilepsy
* Shift working or have a history of shift work within the previous six months
* Currently, or within the previous 8 weeks, consuming any prebiotic or probiotic products/supplements (including specifically oligosaccharides)
* Participation in any other intervention research trials
* Sleeping at a location other than their usual residence more than two nights per week during participation
* Travel across multiple time zones within the last three months or have planned travel across multiple time zones during the study
* Current or recent mood disturbances or Axis I disorders (descriptions will be given)
* Current misuse of alcohol and/or drugs
* Current smoker
* Recent (within the last 12 weeks) infection and/or use of antibiotic medication
* Pregnant, seeking to become pregnant or lactating
* Those using (including within the last 2 weeks) proton-pump inhibitors

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency (SE) | Change from Baseline to end of supplementation period at 28 days
  Sleep efficiency (SE), commonly defined as the ratio of total sleep time (TST) to time in bed (TIB), will be reported as a percentage of time in bed. This data will be obtained from SleepScore analysis. The SleepScore Max (SleepScore Labs, Carlsbad, CA, USA; Sleep Tracker: How The SleepScore Max Works | Sleep.ai) is a non-contact sleep monitoring device designed for bedside use. It measures movement, breathing, and environmental factors such as light and temperature to assess sleep quality and duration. Results are presented as a personalised SleepScore™, accessible via a companion app that offers evidence-based guidance for improving sleep.

SECONDARY OUTCOMES:
Actigraphy - Sleep onset latency | Change from baseline following 28 days of supplement consumption
  recorded minutes taken from intention to sleep to sleep initiation
Actigraphy - Sleep efficiency | Change from baseline following 28 days of supplement consumption
  ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed (percentage)
Actigraphy - Number of awakenings | Change from baseline following 28 days of supplement consumption
  recorded number of awakenings during entire sleep period
Actigraphy - Wake after sleep onset (WASO) | Change from baseline following 28 days of supplement consumption
  recorded minutes awake during the entire sleep period following sleep onset
COMPASS global performance measures | Change from baseline following 28 days of supplement consumption
  Speed of performance, and accuracy of performance measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline following 28 days of supplement consumption
  Pittsburgh Sleep Quality Index (PSQI): Total Score. The PSQI is a validated self-rating instrument assessing aspects of sleep quality.Minimum score 0 (better); maximum score 21 (worse) < or = 5 associated with good sleep quality; > 5 associated with poor sleep quality.
Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | Change from baseline following 28 days of supplement consumption
  A 21-item measure of mood over the previous week (each item is rated on scale from 0-3). Scoring creates 3 component scores: depression, anxiety and stress (each on a scale of 0-21) with higher scores indicating higher symptomology. Cut-off scores, according to each set of symptoms, are available (normal, mild, moderate, severe and extremely severe) or total scores can be derived by multiplying the sum of all three component scores by 2.
State-Trait Anxiety Inventory (STAI) | Change from baseline following 28 days of supplement consumption
  A 40-item measure of current and general anxiety levels. Each item is rated on a scale from 1-4. Scoring creates two components: state anxiety (20 items) and trait anxiety (20 items), with a range for each between 20-80. Following transformation through reversed coding, higher scores indicate higher levels of anxiety
Actigraphy - Total sleep time | Change from baseline following 28 days of supplement consumption
  recorded minutes asleep over entire sleep period
Sleep Diary - Total sleep time | Change from baseline following 28 days of supplement consumption
  recorded minutes asleep over entire sleep period
Sleep Diary - Sleep onset latency | Change from baseline following 28 days of supplement consumption
  logged minutes taken from intention to sleep to sleep initiation
Sleep Diary - Sleep efficiency | Change from baseline following 28 days of supplement consumption
  ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed (percentage)
Sleep Diary - Number of awakenings | Change from baseline following 28 days of supplement consumption
  logged number of awakenings during entire sleep period
Sleep Diary - Wake after sleep onset (WASO) | Change from baseline following 28 days of supplement consumption
  logged minutes awake during the entire sleep period following sleep onset

CONTACTS AND LOCATIONS:
Overall Officials: Professor Jason Ellis, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University- Northumbria Sleep center and NUTRAN, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No